CLINICAL TRIAL: NCT06558422
Title: Human Models of Selective Insulin Resistance: Pancreatic Clamp
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: University of California, Berkeley (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AAAU9702; P30DK063608 (NIH); K12DK133995 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Insulin Resistance; Hyperinsulinemia; Metabolic Dysfunction Associated Steatotic Liver Disease; Non-Alcoholic Fatty Liver Disease; Prediabetic State; Obesity
Keywords: Insulin resistance; Hyperinsulinemia; Diabetes; Non-alcoholic fatty liver disease; Metabolic dysfunction associated steatotic liver disease
MeSH Terms: conditions — Insulin Resistance; Hyperinsulinism; Non-alcoholic Fatty Liver Disease; Prediabetic State; Obesity; Diabetes Mellitus | interventions — Insulin; Octreotide; Glucagon; Human Growth Hormone; Glucose

STUDY DESIGN:
Intervention Model Description: All participants will undergo (i.e., cross over between) both pancreatic clamp protocols (MH, RE) separated by 2-8 weeks. The order of the clamp protocols (i.e., MH > RE, RE > MH) will be randomized.
Who Masked: Participant
Masking Description: Participant will be blinded to study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Maintenance hyperinsulinemia (MH) Protocol then Reduction toward Euinsulinemia (RE) Protocol (Experimental): On Pancreatic Clamp Visit 1 (MH Protocol), the insulin infusion rate (IIR) will be set to approximately replicate participants' endogenous fasting serum insulin levels based on screening visit data for the duration of the pancreatic clamp. On Pancreatic Clamp Visit 2 (RE Protocol), the IIR will be set to reduce serum insulin levels to roughly 50% of the screening fasting serum insulin for the duration of the pancreatic clamp. In both cases, plasma glucose will be clamped to approximately 140 mg/dL +/- 10%.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Growth Hormone, Human; Drug: 20% D-glucose (aq); Diagnostic Test: [6,6-2H2] D-glucose; Diagnostic Test: [1-13C1] sodium acetate; Dietary Supplement: Nestle BOOST Plus; Dietary Supplement: KIND Bar; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer
- Reduction toward euinsulinemia (RE) protocol (Experimental): On Pancreatic Clamp Visit 1 (RE Protocol), the insulin infusion rate (IIR) will be set to produce serum insulin levels of approximately 50% that of the screening fasting serum insulin level for the full duration of the pancreatic clamp. On Pancreatic Clamp Visit 2 (MH Protocol), the IIR will be set to approximately replicate the full fasting serum insulin for the duration of the pancreatic clamp. In both cases, plasma glucose will be clamped to approximately 140 mg/dL +/- 10%.
  Interventions: Drug: Insulin human; Drug: Octreotide Acetate; Drug: Glucagon; Drug: Growth Hormone, Human; Drug: 20% D-glucose (aq); Diagnostic Test: [6,6-2H2] D-glucose; Diagnostic Test: [1-13C1] sodium acetate; Dietary Supplement: Nestle BOOST Plus; Dietary Supplement: KIND Bar; Device: Harvard Apparatus PHD ULTRA CP syringe pump; Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer

INTERVENTIONS:
Drug: Insulin human — Insulin infusion rate (IIR) will be determined either to maintain fasting serum insulin levels (MH protocol) or to reduce fasting serum insulin levels by approximately 50% toward euinsulinemia (RE protocol).
  Other Names: Novolin-R, Humulin-R
Drug: Octreotide Acetate — Octreotide will be infused at 30 ng/kg/min to suppress endogenous insulin, glucagon, and growth hormone secretion. Co-administered with glucagon and rhGH.
Drug: Glucagon — Glucagon will be replaced at a constant rate of up to 0.65 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and rhGH.
Drug: Growth Hormone, Human — Recombinant human growth hormone (rhGH) will be replaced at a constant rate of up to 3 ng/kg/min to maintain baseline counterregulatory response. Co-administered with octreotide and glucagon.
  Other Names: Omnitrope, Zomacton
Drug: 20% D-glucose (aq) — 20% D-glucose (aq) (D20W) will be administered to counteract hypoglycemia or strongly downward blood glucose trends, as needed.
  Other Names: D20W
Diagnostic Test: [6,6-2H2] D-glucose — Stable isotope tracer administered to calculate glucose kinetics during pancreatic clamp.
  Other Names: D2-glucose, D2G
Diagnostic Test: [1-13C1] sodium acetate — Stable isotope tracer administered to calculate de novo lipogenesis during pancreatic clamp.
  Other Names: 13C-acetate, C13A
Dietary Supplement: Nestle BOOST Plus — Nutritional supplement will be administered to provide standardized "mixed meals" prior to the pancreatic clamp.
Dietary Supplement: KIND Bar — Energy bar snack will be administered the evening before the pancreatic clamp.
Device: Harvard Apparatus PHD ULTRA CP syringe pump — Syringe pump used for highly precise administration of insulin, octreotide/glucagon/rhGH, and D20W (as needed) even at low infusion rates.
Device: Yellow Springs Instruments (YSI) 2500 Biochemistry Glucose/Lactate Analyzer — Glucose oxidase analyzer used to detect plasma glucose levels at the point of care. YSI have been the gold standard in clamp studies for many years. Two machines will run in parallel to ensure accuracy of results.

SUMMARY:
This is a single-center, prospective, randomized, controlled (crossover) clinical study designed to investigate the impact of lowering insulin levels on hepatic glucose production (HGP) vs de novo lipogenesis (DNL) in people with insulin resistance. The investigators will recruit participants with a history of overweight/obesity and evidence of insulin resistance (i.e., fasting hyperinsulinemia plus prediabetes and/or impaired fasting glucose and/or Homeostasis Model Assessment of Insulin Resistance [HOMA-IR] score >=2.73), and with evidence of metabolic dysfunction-associated steatotic liver disease (MASLD). Participants will undergo two pancreatic clamp procedures -- one in which serum insulin levels are maintained near hyperinsulinemic baseline (Maintenance Hyperinsulinemia or "MH" Protocol) and the other in which serum insulin levels are lowered by 50% (Reduction toward Euinsulinemia or "RE" Protocol). In both clamps the investigators will use stable-isotope tracers to monitor hepatic glucose and triglyceride metabolism. The primary outcome will be the impact of steady-state clamp insulinemia on HGP vs DNL.

DETAILED DESCRIPTION:
Although high blood sugar and risk of heart disease are the most well-known health effects of type 2 diabetes (T2DM), metabolic dysfunction-associated steatotic liver disease (MASLD), in which too much fat accumulates in the liver, has come to be recognized as another important complication. Unchecked, MASLD can progress to severe liver inflammation, liver failure, and even liver cancer. The investigators suspect that high levels of the blood sugar-lowering hormone insulin leads to excessive fat production by the liver, and so lowering insulin levels might help to improve MASLD. In order to answer this question, the investigators will recruit people with MASLD at risk for T2DM to perform a "pancreatic clamp" - a procedure in which the body's production of insulin is temporarily shut off and then replaced at the same or lower levels. Again, the investigators expect that lowering insulin levels will lower fat production ("de novo lipogenesis" or DNL). Research participants in this prospective, randomized, controlled (crossover) study will therefore undergo two pancreatic clamps in random order: one roughly maintaining their own internal ("basal") insulin level ("MH Protocol") and one in which the investigators lower that basal insulin level by 50% ("RE Protocol"). In each case, the investigators will observe the absolute and relative changes in the liver's production of glucose (hepatic glucose production, HGP) and of triglycerides (de novo lipogenesis, DNL) using stable-isotope tracers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 18-65 years
* Body mass index of 27-50 kg/m2
* Able to understand written and spoken English and/or Spanish
* Evidence of insulin resistance, represented by any or all of the following criteria:

  * Meeting either of the American Diabetes Association's definitions for prediabetes or Impaired fasting glucose (IFG) within the previous year and on screening labs:

    1. Prediabetes: Hemoglobin A1c 5.7-6.4%
    2. IFG: plasma glucose of 100-125 mg/dL after 8-h fast
* Homeostasis Model of Insulin Resistance (HOMA-IR) score ≥ 2.73
* Fasting hyperinsulinemia (fasting insulin level ≥ 13 µU/mL) on screening labs
* Presence of uncomplicated MASLD, defined by vibration-controlled transient elastography (VCTE) as a steatosis score S1-S3 + fibrosis score F0-F2
* Written informed consent (in English or Spanish) and any locally required authorization (e.g., Health Insurance Portability and Accountability Act) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

* Unable to provide informed consent in English or Spanish
* Unwillingness to use only bedpan or urinal to void or to refrain from non-emergent mobile device use during the clamp
* Documented weight loss of ≥ 5% of baseline within the previous 3 months
* Abnormal blood pressure (including on treatment, if prescribed)

  * Systolic blood pressure < 90 mm Hg or > 160 mm Hg, and/or
  * Diastolic blood pressure < 60 mm Hg or > 100 mm Hg
* Abnormal resting heart rate: < 60 or ≥ 110 bpm

  * Sinus brady- or tachycardia that has been worked up and considered benign by the recruit's personal physician may be permitted at the PI's discretion
* Abnormal screening electrocardiogram (or if on file, performed within previous 90 days)
* Laboratory evidence of diabetes mellitus:

  * Hemoglobin A1c ≥ 6.5%, and/or
  * Fasting plasma glucose ≥ 126 mg/dL
* Positive qualitative β-hCG (Human chorionic gonadotropin, β subunit) (i.e., pregnancy test) in women of childbearing potential
* Positive urine drug screen, except for lawfully prescribed medications and/or marijuana
* Liver function abnormalities (either of the following)

  * Transaminases (AST or ALT) > 3.0 x the upper limit of normal
  * Total bilirubin > 1.25 x the upper limit of normal
* Fasting serum triglycerides at screening ≥ 400 mg/dL
* Abnormal screening serum electrolytes that are considered potentially significant according to the clinical judgment of the PI
* Abnormal complete blood count (CBC) (any of the following)

  * Hemoglobin < 10 g/dL or hematocrit < 30%
  * Platelet count < 100,000/µL
* Women currently pregnant, measured by serum and/or urine β-hCG, or trying to become pregnant
* Women currently breastfeeding
* History of having met any of the American Diabetes Association's definitions of diabetes mellitus (i.e., overt diabetes):

  * Hemoglobin A1c ≥ 6.5%, or rapid rise in documented HbA1c values causing clinical concern for evolving insulin deficiency
  * Plasma glucose ≥ 126 mg/dL after 8-h fast
  * Plasma glucose of ≥ 200 mg/dL at 2 h after ingestion of a 75-g glucose load
  * Random plasma glucose ≥ 200 mg/dL associated with typical hyperglycemic symptoms, diabetic ketoacidosis, or hyperglycemic-hyperosmolar state
* History of gestational diabetes mellitus within the previous 5 years
* Use of most antidiabetic medications within the 30 days prior to screening

  * Excluded: thiazolidinediones, sulfonylureas, meglitinides, DPP4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors, amylin mimetics, acarbose, insulin
  * Metformin is acceptable provided that recruits meet all of the inclusion criteria at screening
* Clinical concern for absolute insulin deficiency (e.g., type 1 diabetes, pancreatic disease)
* Known diagnoses of familial combined hyperlipidemia or familial chylomicronemia syndrome
* Use of certain lipid-lowering drugs within 30 d prior to screening visit:

  * Fibrates (e.g., fenofibrate, clofibrate, gemfibrozil)
  * Prescription-strength omega-3 fatty acids (e.g., Lovaza®, Vascepa®)
* Known, documented history, at the time of screening, of any of the following medical conditions:

  * Pancreatic pathology
  * Cardiovascular diseases (N.B. uncomplicated hypertension is not exclusionary)
  * Chronic kidney disease, Stage 3 or higher (estimated glomerular filtration rate < 60 mL min-1 1.73 m-2), of any cause
  * Advanced or severe liver disease (including fibrosis scores of F3-F4 on screening VCTE)
  * Gallstone disease
  * Chronic viral illness
  * Malabsorptive conditions (active)
  * Active seizure disorder (including controlled with antiepileptic drugs)
  * Psychiatric diseases causing functional impairment and/or requiring use of anti-dopaminergic antipsychotic drugs associated with significant weight gain/metabolic dysfunction (e.g., clozapine, olanzapine), monoamine oxidase inhibitors, tricyclic antidepressants, or lithium
  * Known adrenal disease
  * Venous thromboembolic disease (deep vein thrombosis or pulmonary embolism) or any required use of therapeutic anticoagulation
  * Bleeding disorders, including due to anticoagulation, or significant anemia (see above)
  * Active malignancy, or hormonally active benign neoplasm
* Clinical concern for increased risk of volume overload, including due to medications and/or heart/liver/kidney problems, as listed above
* Clinical concern for increased risk of hypokalemia, including low potassium on screening labs (i.e., below lower limit of normal), use of certain medications, or any medical conditions listed above
* Use of certain medications currently or within 30 d prior to screening:

  * Prescribed medications used for any of the indications in the preceding list of excluded conditions, or their use within 30 d prior to screening, except allowances for:
  * Use of drugs prescribed for indications other than the exclusionary diagnoses/purposes listed above, e.g., antiepileptic drugs used for non-seizure indications, ACEi (angiotensin-converting enzyme inhibitor) / ARB (angiotensin receptor blocker) used for uncomplicated hypertension rather than for congestive heart failure, etc. Note, as above, that antidiabetic drugs except metformin within 30 days of screening are excluded.
  * Loop diuretics (furosemide, torsemide, ethacrynic acid)
  * Oral or parenteral corticosteroids (at greater than prednisone 5 mg daily, or equivalent) for more than 3 days within the previous 30 days; topical and inhaled formulations are permitted
  * Fludrocortisone
  * Beta blockers or non-dihydropyridine calcium channel blockers (verapamil or diltiazem)
* History of certain weight-loss (bariatric) surgery, including:

  * Roux-en-Y gastric bypass
  * Biliopancreatic diversion
  * Restrictive procedures (lap band, sleeve gastrectomy) performed within the past 6 months
* Clinical concern for alcohol overuse, including recent documented history during screening and/or participant report of regularly consuming more than 2 drinks per day for males or 1 drink per day for females.
* Positive urine drug screen, with exceptions for:

  * Lawfully prescribed medications
  * Marijuana/THC positivity, provided that the participant agrees not to use it during the same period that they will abstain from alcohol
* History of severe infection or ongoing febrile illness within 14 days of screening
* Any other disease, condition, or laboratory value that, in the opinion of the investigator, would place the participant at an unacceptable risk and/or interfere with the analysis of study data.
* Known allergy/hypersensitivity to any component of the medicinal product formulations, foods (including soy, dairy, peanuts, tree nuts, or egg), IV infusion equipment, plastics, adhesive or silicone, history of infusion site reactions with IV administration of other medicines, or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
* Concurrent enrollment in another clinical study of any investigational drug therapy within 30 days prior to screening or within 5 half-lives of an investigational agent, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2027-01-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Hepatic de novo lipogenesis (DNL) (absolute value) | Up to 6.5 hours of pancreatic clamp protocol
  Percent incorporation of newly synthesized fatty acids into plasma or very low-density lipoprotein (VLDL) triglyceride (TG) during pancreatic clamp procedures. (Unit: %)
Hepatic de novo lipogenesis (DNL) (relative value) | Up to 6.5 hours of pancreatic clamp protocol
  Percent incorporation of newly synthesized fatty acids into plasma or VLDL TG during pancreatic clamp procedures. (Unit: fold difference and/or ∆% versus other group)
Endogenous glucose production (EGP) (absolute value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: mg/kg/min)
Endogenous glucose production (EGP) (relative value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: fold difference and/or ∆% versus other group)
Plasma glucose level | Up to 6.5 hours of pancreatic clamp protocol
  Plasma glucose level during pancreatic clamp procedures. (Units: mg/dL)
Serum insulin level | Up to 6.5 hours of pancreatic clamp protocol
  Serum insulin level during pancreatic clamp procedures (Units: µU/mL)

SECONDARY OUTCOMES:
Serum or plasma triglyceride level | Up to 6.5 hours of pancreatic clamp protocol
  Serum or plasma triglyceride level in response to pancreatic clamp procedures (Units: mg/dL)
Plasma free fatty acids level | Up to 6.5 hours of pancreatic clamp protocol
  Plasma free fatty acids level in response to pancreatic clamp procedures. (Units: mmol/L)
Glucose kinetics: rate of appearance (absolute value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: mg/kg/min)
Glucose kinetics: rate of appearance (relative value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: fold difference and/or ∆% versus other group)
Glucose kinetics: rate of disappearance (absolute value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: mg/kg/min)
Glucose kinetics: rate of disappearance (relative value) | Up to 6.5 hours of pancreatic clamp protocol
  Calculated from D2G tracer enrichment by the Steele equations during pancreatic clamp procedures. (Units: fold difference and/or ∆% versus other group)

OTHER OUTCOMES:
Serum C-peptide level | Up to 6.5 hours of pancreatic clamp protocol
  Serum C-peptide level in response to octreotide infusion during pancreatic clamps. (Units: ng/mL)
Plasma glucagon level | Up to 6.5 hours of pancreatic clamp protocol
  Plasma glucagon level in response to octreotide infusion during pancreatic clamps. (Units: ng/L)
Serum growth hormone level | Up to 6.5 hours of pancreatic clamp protocol
  Serum growth hormone level in response to octreotide infusion during pancreatic clamps. (Units: ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Cook, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Participant-level clinical data will be preserved by depositing the deidentified data to Dryad, a generalist repository that is participating in the NIH Generalist Repository Ecosystem Initiative. The repository will provide metadata, persistent identifiers, and long-term access for open and controlled access. Each study created in Dryad is assigned a digital object identifier (DOI). This data DOI will be referenced in the publication to allow the research community easy access to the exact data used in the publication.
  To protect research participants' privacy and confidentiality, data submitted to the repository will not include personally identifiable information such as names or addresses. Additional protections, such as the approach for managing Health Insurance Portability and Accountability Act identifiers, will be used for de-identification and to provide a limited data set to minimize the risk of participant reidentification.
Time Frame: Scientific data will be shared as soon as possible. Scientific data included in published manuscripts will be available at the time of publication; all other generated scientific data will be shared no later than the end of the award. The study data will be stored in the repository for at least 5 years.
Access Criteria: To request access of the data, researchers will use the standard processes at Dryad. Given that we seek the widest possible availability, in most cases all that is necessary is obtaining a Dryad account from the repository web site.